CLINICAL TRIAL: NCT04320758
Title: One Year Clinical Evaluation of Translucent Zirconia Crowns in Dental Esthetic Zone With Biologically Oriented Preparation Technique (BOPT) Versus Conventional Preparation (Randomized Clinical Trial)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Kareem Talaat Abdelwahab Ahmed Ali, Resident,Fixed Prosthodontics Department,Faculty of Dentistry, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019-09-30
Record Dates: First submitted 2020-03-23; First posted 2020-03-25 (Actual); Last update posted 2020-09-17 (Actual); Status verified 2020-09

CONDITIONS: Single Crowns in Aesthetic Dental Zone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- single crown in dental aesthetic zone (Experimental): teeth in dental aesthetic zone
  Interventions: Other: conventional preparation design
- teeth need single crown in dental aesthetic zone (Experimental): teeth in dental aesthetic zone
  Interventions: Other: biologically oriented preparation technique

INTERVENTIONS:
Other: conventional preparation design — chamfer finish line
  Other Names: horizontal preparation technique
  Arms: single crown in dental aesthetic zone
Other: biologically oriented preparation technique — shoulder less preparation design
  Other Names: vertical perpetration technique
  Arms: teeth need single crown in dental aesthetic zone

SUMMARY:
Aim of the studyto evaluate the clinical behavior of translucent zirconia crown in dental esthetic zone with biologically oriented preparation technique versus conventional preparation.

ELIGIBILITY:
Inclusion Criteria:

* All subjects are required to be:

  1. From 21-35 years old, be able to read and sign the informed consent document.
  2. Have no active periodontal or pulpal diseases, have teeth with good restorations
  3. Psychologically and physically able to withstand conventional dental procedures
  4. Patients with teeth problems indicated for single all ceramic restoration in maxillary esthetic zone cr

     1. Badly decayed teeth
     2. Teeth restored with large filling restorations
     3. Endodontically treated teeth
     4. Malformed teeth
     5. Malposed teeth (Tilted, over-erupted, rotated, etc.)
     6. Spacing between maxillary teeth in esthetic zone
  5. Able to return for follow-up examinations and evaluation

Exclusion Criteria:

1. Patient less than 21or more than 35 years
2. Patient with active resistant periodontal diseases
3. Patients with poor oral hygiene and uncooperative patients
4. Pregnant women
5. Patients in the growth stage with partially erupted teeth
6. Psychiatric problems or unrealistic expectations
7. Patient with periodontal problems
8. patients with malocclusion or parafunctional habits

Ages: 21 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 22 (Estimated)
Dates: Start 2020-10-30 (Estimated); Primary Completion 2020-10-30 (Estimated); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
Marginal adaptation | 1 year
  Measured using Modified USPHS criteria1

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of dentistry Cairo university, Cairo, New Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided